CLINICAL TRIAL: NCT06254781
Title: Luspatercept in Metastatic Adult Granulosa Cell Tumor (AGCT) of the Ovary
Brief Title: Luspatercept in Metastatic AGCT of the Ovary
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OZUHN-015; 22-5326 (Other: University Health Network)
Record Dates: First submitted 2022-05-26; First posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Adult Granulosa Cell Tumor of the Ovary
MeSH Terms: conditions — Granulosa cell tumor of the ovary | interventions — luspatercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Luspatercept in metastatic AGCT of the ovary (Experimental): Luspatercept, 1.0 mg/kg, subcutaneously, every three weeks
  Interventions: Drug: Luspatercept

INTERVENTIONS:
Drug: Luspatercept — Erythroid Maturation Agent
  Other Names: Reblozyl

SUMMARY:
This is a single participant study of luspatercept for the treatment of a patient with dult granulosa cell tumor (AGCT) of the ovary.

DETAILED DESCRIPTION:
This patient has AGCT driven by a somatic oncogenic FOXL2 mutation identified through a molecular profiling study. One of the ways in which this mutation drives tumorigenesis is via increased activity of SMAD3, which results in decreased expression of follistatin and allows increased signalling of activin, a TGFB ligand that activates the TGFB pathway. Anti-TGFB approaches have shown promise in preclinical studies of AGCTs and several early phase trials are investigating different levels of TGFB pathway inhibition1.

As an activin receptor ligand trap, luspatercept has been shown to reduce SMAD2/3 signaling and improve anemia in disorders characterized by ineffective erythropoiesis, such as B-thalassemia and myelodysplastic syndromes (MDSs). This study aims to determine if we can apply this rationale to a patient with recurrent AGCT with oncogenic FOXL2 mutation known to drive TGFB/SMAD pathway overactivity.

Luspatercept has not been investigated in AGCT and therefore the efficacy of this specific agent as a cancer therapeutic is not yet known. Other TFGB ligand-trapping agents are in development and early phase clinical trials. One such example is AVID200, a TGFB ligand trap and selective inhibitor of TGFB1 and advanced solid tumors. There were 19 patients included in a phase I study of AVID200 monotherapy in patients with advanced solid tumors. A best response of stable disease for over 12 weeks seen in two patients (adenoid cystic carcinoma and breast carcinoma). The maximum tolerated dose was not reached; no Grade 3 adverse events were seen and only three adverse events were reported overall including diarrhea and lipase elevation.

ELIGIBILITY:
Inclusion Criteria:

* N/A

Exclusion Criteria:

* N/A

This patient's case was recently discussed in the hospital expert molecular tumor board rounds consisting of representatives from specialist genomic profiling and gynecologic medical oncology departments. The discussion surrounded the best next therapeutic option in this rare cancer subtype without clear standard of care guidelines. The recommendation from this discussion was to investigate targets of the TGFβ pathway, such as luspatercept. Therefore, specific eligibility criteria aside from individual patient's medical history is not applicable.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-05-30 (Actual); Primary Completion 2022-08-22 (Actual); Study Completion 2022-08-29 (Actual)

PRIMARY OUTCOMES:
Objective response | From baseline CT until disease progression or until the investigator deems that it is in the patient's best interest to stop study treatment, whichever came first, assessed up to 3 months.
  By computed tomography (CT) scans
Eastern Cooperative Oncology Group (ECOG) score | From baseline ECOG until disease progression or until the investigator deems that it is in the patient's best interest to stop study treatment, whichever came first, assessed up to 3 months.
  0. Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  3. Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  4. Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  5. Death
Circulating tumor DNA (ctDNA) levels | From baseline ctDNA until disease progression or until the investigator deems that it is in the patient's best interest to stop study treatment whichever came first, assessed up to 3 months..
  Observe change between baseline ctDNA until disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Amit Oza, M.D., Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada